CLINICAL TRIAL: NCT03218592
Title: ENLIGHTEN: Establishing Novel Antiretroviral (ARV) Imaging for Hair to Elucidate Non-Adherence
Acronym: ENLIGHTEN
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: 17-0546; 1R01AI122319-01 (NIH)
Record Dates: First submitted 2017-07-10; First posted 2017-07-14 (Actual); Results first posted 2019-11-22 (Actual); Last update posted 2019-11-22 (Actual); Status verified 2019-02

CONDITIONS: HIV/AIDS
Keywords: Adherence; Hair
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Maraviroc; dolutegravir; Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination; Tenofovir; Emtricitabine

STUDY DESIGN:
Intervention Model Description: Prospective. Single-center, open-label, 3-arm, triple stage study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Maraviroc (Experimental): 12 Healthy subjects will dose with Maraviroc Pill and we will collect blood and hair over all three phases
  Interventions: Drug: Maraviroc Pill
- Dolutegravir (Experimental): 12 Healthy volunteers will dose with Dolutegravir Pill and we will collect blood and hair over all three phases
  Interventions: Drug: Dolutegravir Pill
- Truvada (Experimental): 12 healthy volunteers will dose with Truvada Pill and we will collect blood and hair over all three phases
  Interventions: Drug: Truvada Pill

INTERVENTIONS:
Drug: Maraviroc Pill — Subjects will take a single dose in Phase 1, Daily Doses in Phase 2 for 28 days, and then be randomized in Phase 3 to zero doses, one dose a week or three doses weekly
  Other Names: selzentry
  Arms: Maraviroc
Drug: Dolutegravir Pill — Subjects will take a single dose in Phase 1, Daily Doses in Phase 2 for 28 days, and then be randomized in Phase 3 to zero doses, one dose a week or three doses weekly
  Other Names: Tivicay
  Arms: Dolutegravir
Drug: Truvada Pill — Subjects will take a single dose in Phase 1, Daily Doses in Phase 2 for 28 days, and then be randomized in Phase 3 to zero doses, one dose a week or three doses weeklySubjects will take a single dose in Phase 1, Daily Doses in Phase 2 for 28 days, and then be randomized in Phase 3 to zero doses, one dose a week or three doses weekly
  Other Names: Tenofovir/Emtricitabine
  Arms: Truvada

SUMMARY:
Purpose: Perform a 3-phase (single dose, multi dose, dose proportionality) study in healthy volunteers using daily tenofovir+emtricitabine, dolutegravir, and maraviroc dosing to quantify intra- and inter-subject variability and dose proportionality. The influence of covariates on ARV hair distribution (e.g., hair growth rate, race, hair color, hair treatment) will also be measured. Using both population PK modeling and physiologic based PK (PBPK) approaches, a statistical model to quantify ARV adherence patterns based on signal intensity/pattern will be developed.

Participants: Healthy volunteers, aged 18 to 70 years of age, inclusive on the date of screening, with an intact gastrointestinal system and at least 1cm caput hair.

Procedures (methods): Participants will be sequentially assigned to enroll in a dosing arm, beginning with maraviroc (MVC), then dolutegravir (DTG), and ending with tenofovir/emtricitabine (TFV/FTC). All participants will take a single observed dose of study product in Phase 1, with blood and hair samples obtained on Days 3, 7, 14, 21 and 28 days post-dose. In Phase 2, all participants take 28 days straight of daily dosing, observed, of the same study product. Blood and hair samples obtained on the same days post-dose. In Phase 3, participants will be randomized to stop their drug, or decrease dosing to one or three doses weekly. Hair and blood samples will again be obtained on the same days post-dose. All participants will complete a follow-up safety visit with 14 days of completing study sampling.

DETAILED DESCRIPTION:
Details:

Participants will be sequentially assigned to enroll in dosing arm, beginning with Maraviroc, then Dolutegravir and ending with Tenofovir/Emtricitabine, Participation will last approximately 3 months and will include a screening visit, three 28-day phases, and a follow-up safety visit.

Phase 1 consists of a 28-day study period with a single dose of study product on Day 0.

Phase 2 consists of a 28-day study period with each subject receiving a single daily observed dose of study product beginning on Day 0.

Phase 3 consists of a 28-day study period, with three randomized drug-dosing schemas beginning on Day 0. Participants will either: stop taking their study product, dose once per week, or dose three times per week.

Participants will return to the clinic for hair and blood sampling on days 3/7/14/21/28 post-dose for all three phases. Adverse events will be assessed at every visit. Safety labs will be drawn at the midpoint and at the end of each study phase, and at any time indicated due to suspected adverse events.

Description of Study Phases Screening: Participants will be recruited from a variety of advertisements, and pre-screened using a telephone Institutional Review Board (IRB)-approved questionnaire. If participants are interested and pass the initial screening, a screening study visit in the research center will be scheduled. This visit should take approximately 90 minutes, during which full physical examination and medical history will be obtained, as well as physical diagnostics to assess for eligibility. This visit must be completed within the 28 days prior to enrollment.

Phase 1: Consists of a 28-day study period, with a single dose of study product on Day 0 (Maraviroc, Dolutegravir, or tenofovir/emtricitabine). Day 0 can be scheduled on either Mondays or Tuesdays, and once eligibility is confirmed on the day of enrollment, a witnessed dose of study product will be administered. Participants will return to the clinic for hair and blood sampling on Days 3/7/14/21/28 days post-dose. Adverse events will be assessed at every visit. Safety labs will be drawn at the midpoint and at the end of the study phase, and at any time indicated due to suspected adverse events. These visits should last less than 30 minutes.

Phase 2: Consists of a 28-day study period, with each subject receiving a single daily observed dose of study product beginning on Day 0. Day 0 can be scheduled on either Mondays or Tuesdays, once continued eligibility is confirmed. Target scheduling will have Phase 2 begin within 2 weeks of completing Phase 1, but could be extended up to 28 days as clinic availability dictates. Participants will return to the clinic daily for dosing, and for hair and blood sampling on Days 3/7/14/21/28 days post-dose. Adverse events will be assessed at every visit. Safety labs will be drawn at the midpoint, and at the end of the study phase, and at any time indicated due to adverse events. These visits should last less than 30 minutes. Dosing only visits should last less than 5 minutes.

Phase 3: Consists of a 28-day study period, with three randomized drug-dosing schemas. Day 0 can be scheduled on Mondays, Tuesdays or Fridays, once continued eligibility is confirmed. Target scheduling will have Phase 3 begin as soon as possible after completing Phase 2, on a Monday/Tuesday/Or Friday within the week. On Day 0, participants will be randomized to one of 3 potential dosing schemes:

1. No further doses
2. One dose weekly (Day 0, 7, 14, 21) 4 doses
3. Three Doses weekly (Mondays, Wednesdays, Fridays) (Days 0, 2, 4, 7, 9, 11, 14, 16, 18, 21, 23, 25) 12 doses

Participants will return to clinic for observed dosing as scheduled, and for hair and blood sampling on days 3/7/14/21/28). Safety labs will be drawn at the midpoint, at the end, and at any time indicated due to adverse events. These visits should last less than 30 minutes. Dosing only visits should last less than five minutes.

ELIGIBILITY:
Inclusion Criteria

* Healthy volunteer between the ages of 18 and 70, inclusive on the date of screening, with an intact gastrointestinal tract. Healthy is defined as no clinically relevant abnormalities identified by a detailed medical history, full physical examination, including blood pressure and pulse rate measurement, and clinical laboratory tests
* Recent medical history in good medical standing, without evidence of fever five days prior to enrollment
* HIV-negative
* Able to swallow pills
* Has minimum hair required to provide study samples
* Not allergic to any component of the study drug
* Signed and dated informed consent indicating that they have been informed of all pertinent details of the trial and are willing to participate
* Willing and able to comply with scheduled visits, laboratory tests and trial procedures
* Willing to use at least one form of acceptable birth control throughout the duration of the study
* Negative, or receiving treatment, for syphilis at screening
* Hemoglobin Grade 2 or lower, with no clinically significant medical issues that would preclude blood sampling

Exclusion Criteria

* Age outside of desired range
* Confirmed positive results for HIV, Hepatitis B or C at screening
* Subjects of all genders actively involved in the conception process, in addition to cisgender female subjects who are in the immediate post-partum period or breastfeeding
* Insufficient amount of hair or unwilling to keep hair length at least 1 centimeter throughout duration of study
* Unable or unwilling to comply with all lifestyle measures and/or visits
* Impaired renal function, as documented by a creatinine clearance <80 mL/min with the Cockcroft-Gault equation
* Has donated blood within the past 56 days in the amount greater than 500 mL
* Has taken an investigational drug in the past 4 months
* Clinical, laboratory, or surgical abnormalities that would preclude sample collection
* Has a condition, which, in the opinion of the investigator, is likely to interfere with follow-up or ability to take the study medication appropriately
* Any clinically significant laboratory result Grade 2 or greater according to the Division of AIDS (DAIDS) Laboratory Grading Tables
* History of regular alcohol consumption exceeding 14 drinks (1 drink = 5 ounces (150 mL) of wine or 12 ounces (360 mL) of beer or 1.5 ounces (45 mL) of spirits) per week

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2017-06-28 (Actual); Primary Completion 2018-12-03 (Actual); Study Completion 2018-12-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Angela DM Kashuba, BScPhmPharmD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- Clinical and Translational Research Center, UNC Hospitals, Chapel Hill, North Carolina, United States

REFERENCES:
- [Derived] Hill LM, Golin CE, Pack A, Carda-Auten J, Wallace DD, Cherkur S, Farel CE, Rosen EP, Gandhi M, Asher Prince HM, Kashuba ADM. Using Real-Time Adherence Feedback to Enhance Communication About Adherence to Antiretroviral Therapy: Patient and Clinician Perspectives. J Assoc Nurses AIDS Care. 2020 Jan-Feb;31(1):25-34. doi: 10.1097/JNC.0000000000000089. PMID 31033629

RESULTS

PARTICIPANT FLOW:
Period: Phase 1: 1 Dose
Arm/Group | Maraviroc | Dolutegravir | Truvada
Started | 12 | 12 | 12
Completed | 12 | 12 | 12
Not Completed | 0 | 0 | 0
Period: Phase 2: Daily Doses x 28 Days
Arm/Group | Maraviroc | Dolutegravir | Truvada
Started | 12 | 12 | 12
Completed | 12 | 12 | 12
Not Completed | 0 | 0 | 0
Period: Phase 3: 0 Doses Per Week
Arm/Group | Maraviroc | Dolutegravir | Truvada
Started | 4 | 4 | 4
4 Patients Per Group | 4 | 4 | 4
Completed | 4 | 4 | 4
Not Completed | 0 | 0 | 0
Period: Phase 3: 1 Dose Per Period
Arm/Group | Maraviroc | Dolutegravir | Truvada
Started | 4 | 4 | 4
4 Patients Per Group | 4 | 4 | 4
Completed | 4 | 4 | 4
Not Completed | 0 | 0 | 0
Period: Phase 3: 3 Doses Per Week
Arm/Group | Maraviroc | Dolutegravir | Truvada
Started | 4 | 4 | 4
4 Patients Per Group | 4 | 4 | 4
Completed | 4 | 4 | 4
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Healthy volunteer adults across all racial, gender and ethnicity spectrums were enrolled. Pregnant or lactating women were excluded.
Groups:
- Truvada: 12 healthy volunteers will dose with Truvada (TFV/FTC) Pill and we will collect blood and hair over all three phases
  Truvada Pill: Subjects will take a single dose in Phase 1, Daily Doses in Phase 2 for 28 days, and then be randomized in Phase 3 to zero doses, one dose a week or three doses weekly. Subjects will take a single dose in Phase 1, Daily Doses in Phase 2 for 28 days, and then be randomized in Phase 3 to zero doses, one dose a week or three doses weekly
- Total: Total of all reporting groups
Arm/Group | Maraviroc | Dolutegravir | Truvada | Total
Number analyzed (Participants) | 12 | 12 | 12 | 36
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 12 | 12 | 12 | 36
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 31 [22.25 to 45] | 42 [30.5 to 51.5] | 26.5 [23.75 to 41.75] | 32 [24.75 to 47]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 9 | 10 | 29
  Male | 2 | 3 | 2 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 0 | 1 | 4
  Not Hispanic or Latino | 9 | 12 | 11 | 32
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 1
  Asian | 1 | 0 | 3 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 1 | 2
  White | 10 | 11 | 8 | 29
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 12 | 12 | 12 | 36
Healthy Volunteer Status [Count of Participants; unit: Participants] | 12 | 12 | 12 | 36

OUTCOME MEASURES:

1. Primary Outcome: Hair Antiretroviral Imaging
Description: Signal Strength concentrations will be measured in hair for all study drugs, inclusive of FTC (emtricitabine), tenofovir (TFV), maraviroc (MRV), and dolutegravir (DTG) using Matrix-assisted Laser Desorption Electrospray Ionization (IR-MALDESI) to be reported by signal abundance (au). Signal abundance is the industry standard unit, and higher values represent greater signal with capability to relate to comparative concentrations.
Time Frame: Up to 28 days post dose
Population: In Phase 3, the 12 participants were divided into 3 dosing categories: either zero further doses,1 dose per week, or 3 doses per week. For the single dose Phase 1, signal abundance was not able to be observed consistently for all drug arms
Measure: Median (Inter-Quartile Range); unit: Signal Abundance (au)
Groups:
- Truvada: 12 healthy volunteers will dose with Truvada Pill and we will collect blood and hair over all three phases
  Truvada Pill: Subjects will take a single dose in Phase 1, Daily Doses in Phase 2 for 28 days, and then be randomized in Phase 3 to zero doses, one dose a week or three doses weekly. Subjects will take a single dose in Phase 1, Daily Doses in Phase 2 for 28 days, and then be randomized in Phase 3 to zero doses, one dose a week or three doses weekly.
Arm/Group | Maraviroc | Dolutegravir | Truvada
Number analyzed (Participants) | 12 | 12 | 12
Signal Abundance (au)
  Phase 3: Zero Doses Per Week: number analyzed (Participants) | 4 | 4 | 4
  Phase 3: Zero Doses Per Week | 156.4826656 [112.6510968 to 180.8064285] | 1092.130868 [688.7225983 to 1325.75008] | 0.501209 [0.2506045 to 11.540693]
  Phase 3: 1 Dose Per week: number analyzed (Participants) | 4 | 4 | 4
  Phase 3: 1 Dose Per week | 3942.692396 [1054.128706 to 7097.7465] | 2377.868226 [1241.605663 to 3519.225695] | 156.1127125 [123.2479595 to 177.8878063]
  Phase 3: 3 Doses Per Week: number analyzed (Participants) | 4 | 4 | 4
  Phase 3: 3 Doses Per Week | 27814.98823 [7059.467332 to 47573.27029] | 5504.883169 [3993.758552 to 6547.002816] | 466.7986895 [416.4048878 to 517.1924913]
  Phase 2: Daily Dosing: number analyzed (Participants) | 4 | 4 | 4
  Phase 2: Daily Dosing | 46013.29104 [14567.14721 to 62292.81721] | 14251.46653 [7003.462543 to 18357.12725] | 824.721385 [593.842582 to 1378.448229]
  Phase 1: Single Dose: number analyzed (Participants) | 4 | 4 | 4
  Phase 1: Single Dose | NA [0 to 0] — For the single dose Phase 1, signal abundance was not able to be observed consistently for all drug arms | NA [0 to 0] — For the single dose Phase 1, signal abundance was not able to be observed consistently for all drug arms | NA [0 to 0] — For the single dose Phase 1, signal abundance was not able to be observed consistently for all drug arms

2. Secondary Outcome: Peripheral Blood Mononuclear Cells (PBMC) Antiretroviral Concentrations
Description: Concentrations of emtricitabine-triphosphate, tenofovir-diphosphate will be measured in peripheral blood mononuclear cells in the Truvada arm only. Truvada is a combination pill, so results for both FTC and TFV are reported in separate columns.
Time Frame: Up to 28 days post-dose
Population: PBMC Concentrations were analyzed in the Truvada arm only. Results are for emtricitabine-triphosphate.
Measure: Median (Inter-Quartile Range); unit: fmol/10^6 cells
Groups:
- Tenfovir (Truvada): 12 healthy volunteers will dose with Truvada Pill and we will collect blood and hair over all three phases
  Truvada Pill: Subjects will take a single dose in Phase 1, Daily Doses in Phase 2 for 28 days, and then be randomized in Phase 3 to zero doses, one dose a week or three doses weeklySubjects will take a single dose in Phase 1, Daily Doses in Phase 2 for 28 days, and then be randomized in Phase 3 to zero doses, one dose a week or three doses weekly
- Emtricitabine (Truvada): 2nd Component in the combo pill Truvada
Arm/Group | Maraviroc | Dolutegravir | Tenfovir (Truvada) | Emtricitabine (Truvada)
Number analyzed (Participants) | 0 | 0 | 12 | 12
fmol/10^6 cells
  Phase 1 Single Dose |  |  | 2.1 [1.2 to 18.5] | 27.09 [1.74 to 465.7]
  Phase 2: 7 Doses per Week |  |  | 127.1 [101 to 185] | 4460 [3620 to 5930]
  Phase 3: 3 Doses Per Week: number analyzed (Participants) | 0 | 0 | 4 | 4
  Phase 3: 3 Doses Per Week |  |  | 60 [54.6 to 71.8] | 2388.69 [1341.4 to 3071.35]
  Phase 3: 1 Dose Per Week: number analyzed (Participants) | 0 | 0 | 4 | 4
  Phase 3: 1 Dose Per Week |  |  | 15.7 [12.2 to 24.2] | 267.82 [194.49 to 453.27]
  Phase 3: Zero Doses per week: number analyzed (Participants) | 0 | 0 | 4 | 4
  Phase 3: Zero Doses per week |  |  | 10.4 [3.5 to 18.5] | 27.48 [1.11 to 135.28]

3. Secondary Outcome: Plasma Antiretroviral Concentrations
Description: Concentrations will be measured in hair of all study drugs, inclusive of FTC (emtricitabine), TFV (tenofovir), MRV (Maraviroc), and DTG (dolutegravir)
Time Frame: Up to 28 days post-dose
Population: 3 drug arms, but Truvada is inclusive of both TFV-dp and FTC-tp
Measure: Median (Inter-Quartile Range); unit: ng/mL
Groups:
- Tenofovir; Emtricitabine: 12 healthy volunteers will dose with Truvada Pill and we will collect blood and hair over all three phases
  Truvada Pill: Subjects will take a single dose in Phase 1, Daily Doses in Phase 2 for 28 days, and then be randomized in Phase 3 to zero doses, one dose a week or three doses weeklySubjects will take a single dose in Phase 1, Daily Doses in Phase 2 for 28 days, and then be randomized in Phase 3 to zero doses, one dose a week or three doses weekly
Arm/Group | Maraviroc | Dolutegravir | Tenofovir | Emtricitabine
Number analyzed (Participants) | 12 | 12 | 12 | 12
ng/mL
  Phase 1: Single dose | 1 [1 to 1] | 1 [1 to 3.455] | 0.5 [0.5 to 0.5] | 0.5 [0.5 to 1.2]
  Phase2: 7 Doses per Week | 9.715 [7.765 to 12.575] | 1240 [797 to 1555] | 61.9 [51.1 to 72.9] | 72.3 [60.3 to 91.4]
  Phase 3: 3 Doses Per Week: number analyzed (Participants) | 4 | 4 | 4 | 4
  Phase 3: 3 Doses Per Week | 1.71 [1.18775 to 3.955] | 69.3 [31.4 to 155] | 9.4 [6.6 to 45.3] | 17.2 [8.8 to 57.8]
  Phase 3: 1 Dose Per Week: number analyzed (Participants) | 4 | 4 | 4 | 4
  Phase 3: 1 Dose Per Week | 1 [1 to 1] | 3.095 [1.4175 to 5.875] | 0.5 [0.5 to 0.7] | 1.2 [0.9 to 1.9]
  Phase 3: 0 Doses per week: number analyzed (Participants) | 4 | 4 | 4 | 4
  Phase 3: 0 Doses per week | 1 [1 to 1] | 1 [1 to 1.2725] | 0.5 [0.5 to 0.5] | 0.5 [0.5 to 0.8]

4. Secondary Outcome: Whole Blood Antiretroviral Concentrations
Description: Concentrations will be measured in dried blood spots of all study drugs, inclusive of FTC (emtricitabine), TFV (tenofovir), MRV (Maraviroc), and DTG (dolutegravir). Truvada is a combination pill, so results for both FTC and TFV are reported in separate columns.
Time Frame: Up to 28 days post-dose
Population: 3 drug arms, but Truvada is inclusive of both TFV/FTC so reported here separately
Measure: Median (Inter-Quartile Range); unit: fmol / 3mm punch
Groups:
- Emtricitabine: 12 healthy volunteers will dose with Truvada Pill and we will collect blood and hair over all three phases
  Truvada Pill: Subjects will take a single dose in Phase 1, Daily Doses in Phase 2 for 28 days, and then be randomized in Phase 3 to zero doses, one dose a week or three doses weekly. Subjects will take a single dose in Phase 1, Daily Doses in Phase 2 for 28 days, and then be randomized in Phase 3 to zero doses, one dose a week or three doses weekly
Arm/Group | Maraviroc | Dolutegravir | Tenofovir | Emtricitabine
Number analyzed (Participants) | 12 | 12 | 12 | 12
fmol / 3mm punch
  Phase 1: Single Dose | 3 [3 to 3] | 10 [10 to 20] | 50 [50 to 50] | 50 [50 to 50]
  Phase 2: 7 Doses per Week | 9.185 [7.76 to 11.625] | 718.5 [482.5 to 937.75] | 809.5 [504.8 to 1107.5] | 280 [214.2 to 345.7]
  Phase 3: 3 Doses Per Week: number analyzed (Participants) | 4 | 4 | 4 | 4
  Phase 3: 3 Doses Per Week | 3 [3 to 4.2025] | 60.95 [39 to 166.75] | 811 [698 to 1027.5] | 150.5 [50 to 221.3]
  Phase 3: 1 Dose Per Week: number analyzed (Participants) | 4 | 4 | 4 | 4
  Phase 3: 1 Dose Per Week | 3 [3 to 3] | 10 [10 to 20] | 644.5 [598.2 to 1007.5] | 50 [50 to 50]
  Phase 3: 0 Doses per week: number analyzed (Participants) | 4 | 4 | 4 | 4
  Phase 3: 0 Doses per week | 3 [3 to 3] | 10 [10 to 12.5] | 621 [433.5 to 906] | 50 [50 to 50]

ADVERSE EVENTS:
Time Frame: 98 days across the individual study period
Description: We have not broken down the AE data per Phase or dosing cohort since there were none to report across any of those groups.
Groups:
- Maraviroc: 12 Healthy subjects will dose with Maraviroc Pill and we will collect blood and hair over all three phases
  Maraviroc Pill: Subjects will take a single dose in Phase 1, Daily Doses in Phase 2 for 28 days, and then be randomized in Phase 3 to zero doses, one dose a week or three doses weekly
  Adverse Events (AEs) reported for participants across all dose groups as there were none to report.
- Dolutegravir: 12 Healthy volunteers will dose with Dolutegravir Pill and we will collect blood and hair over all three phases
  Dolutegravir Pill: Subjects will take a single dose in Phase 1, Daily Doses in Phase 2 for 28 days, and then be randomized in Phase 3 to zero doses, one dose a week or three doses weekly
  AEs reported for participants across all dose groups as there were none to report.
- Truvada: 12 healthy volunteers will dose with Truvada Pill and we will collect blood and hair over all three phases
  Truvada Pill: Subjects will take a single dose in Phase 1, Daily Doses in Phase 2 for 28 days, and then be randomized in Phase 3 to zero doses, one dose a week or three doses weeklySubjects will take a single dose in Phase 1, Daily Doses in Phase 2 for 28 days, and then be randomized in Phase 3 to zero doses, one dose a week or three doses weekly
  AEs reported for participants across all dose groups as there were none to report.
Arm/Group | Maraviroc | Dolutegravir | Truvada
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 0/12 | 0/12 | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-08-24): https://cdn.clinicaltrials.gov/large-docs/92/NCT03218592/Prot_SAP_000.pdf